CLINICAL TRIAL: NCT02425696
Title: Registry of Right-to-left Shunt Detection by Contrast-enhanced Transcranial Doppler in Chinese Population
Status: Completed | Type: Observational
Sponsor: Yingqi Xing (Other)
Responsible Party: Sponsor-Investigator, Yingqi Xing, Director of Head and Neck Vascular Ultrasound Center, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: RLS-1dzx
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2016-10

CONDITIONS: Right-to-left Shunt; Migraine; Cerebral Infarction
Keywords: right-to-left shunt; contrast-enhanced transcranial Doppler; migraine; silent cerebral infarction
MeSH Terms: conditions — Migraine Disorders; Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group 1: Normal individuals without migraine
- group 2: Migraineurs

SUMMARY:
The purpose of the study is to evaluate the prevalence and extent of right-to-left shunt (RLS) in Chinese migraineurs, and the morbidity of silent cerebral infarction in migraineurs.

DETAILED DESCRIPTION:
This is a prospective multicenter study of Chinese population. Participants (normal individuals without migraine and migraineurs) are included after standardized diagnostic procedures (TCD and c-TCD). For migraineurs with large RLS further examinations (c-TTE and brain MRI) are required. Up to 10 study sites nationwide will be needed to recruit the planned participant population during a 1-year period.

The information of each participants will be registered, including basic facts, the longitudinal headache history, frequency, location, quality, intensity, duration, accompanied symptoms, precipitating and exacerbating factors, with or without aura, MIDAS and HIT-6 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* For group 1: Normal healthy individual without migraine.
* For group 2: Clinical history of migraine diagnosed by a neurologist according to the International Classification of Headache Disorders.

Exclusion Criteria:

* Subjects with stenotic intracranial or extracranial arteries or intracranial abnormalities diagnosed with TCD.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We detect RLS through contrast-enhanced transcranial Doppler (c-TCD). The normal individuals will be selected to group 1, while those who suffer from migraine will be selected to group 2. Patients of group 2 with large RLS are required to take TTE and brain MRI.
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
contrast-enhanced transcranial Doppler | 1 year

SECONDARY OUTCOMES:
brain MRI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yingqi Xing, MD, PhD, Study Chair — The First Hospital of Jilin University; Yi Yang, MD, PhD, Study Director — The First Hospital of Jilin University; Yuzhu Guo, Principal Investigator — The First Hospital of Jilin University; Jie Zhang, MD, Principal Investigator — The First Hospital of Jilin University; Sibo Wang, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang XH, Wang SB, Tian Q, Zhong C, Zhang GL, Li YJ, Lin P, You Y, Guo R, Cui YH, Xing YQ. Right-to-left shunt and subclinical ischemic brain lesions in Chinese migraineurs: a multicentre MRI study. BMC Neurol. 2018 Feb 14;18(1):18. doi: 10.1186/s12883-018-1022-7. PMID 29444659